CLINICAL TRIAL: NCT03978494
Title: Randomized, Multicenter, Open-Label, Two-period, Two-sequence Crossover Comparative Pharmacokinetic Study of Generic Tacrolimus (Sandoz) and Advagraf® in Stable Renal Transplant Patients (TODAY)
Brief Title: Study to Compare Pharmacokinetics of Tacrolimus Prolonged-release (PR) Capsules and Advagraf® PR Capsules in Stable Kidney Transplant Patients.
Acronym: TODAY
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: company decision
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1829-TAC-1; 2018-002672-40 (EudraCT Number)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant; Renal transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: Advagraf®; Period 2: Generic tacrolimus (Experimental): In Period 1 patients will receive branded tacrolimus (Advagraf®) orally once-a-day and in Period 2 patients will receive the generic tacrolimus (Sandoz) orally once-a-day.
  Interventions: Drug: Advagraf®; Drug: Generic tacrolimus
- Period 1: Generic tacrolimus; Period 2: Advagraf® (Experimental): In Period 1 patients will receive the generic tacrolimus (Sandoz) orally once-a-day and in Period 2 patients will receive branded tacrolimus (Advagraf®) orally once-a-day.
  Interventions: Drug: Advagraf®; Drug: Generic tacrolimus

INTERVENTIONS:
Drug: Advagraf® — Advagraf®1 mg and 5 mg prolonged-release hard capsules once daily (reference medicinal product).
Drug: Generic tacrolimus — Tacrolimus 1 mg and 5 mg prolonged release hard capsules (Sandoz) once daily (test medicinal product)

SUMMARY:
Study to compare pharmacokinetics of tacrolimus prolonged-release (PR) capsules and Advagraf® PR capsules in stable kidney transplant patients.

DETAILED DESCRIPTION:
Initially, patients will enter a short screening period, and those who continue to meet the inclusion and exclusion criteria will be randomized to receive either test or reference medicinal product in Period 1. In period 2 they will switch to the other formulation. During the whole treatment period four full-pharmacokinetics profiles will be established.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 years;
* Patients with a Body Mass Index (BMI) included in the interval [18.5-33.0] kg/m²;
* Patients who received a primary kidney transplant at least 12 months prior to study entry

Exclusion Criteria:

* Evidence or suspicion of ongoing or persistent, acute or chronic rejection;
* Requirement for dialysis within the six months prior to study entry;
* Glomerular filtration rate (GFR) <30 mL/min
* Pregnant or breastfeeding women, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test;
* Intolerance to tacrolimus, excipients (including lactose, fructose or galactose), or similar products;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2020-05-03 (Estimated); Study Completion 2020-05-03 (Estimated)

PRIMARY OUTCOMES:
AUC(0-τ)ss | Day 21 of each treatment period
  Area under the whole blood concentration curve during a dosage interval (τ=24 hours) at steady state
Cmax,ss | Day 21 of each treatment period
  Maximum whole blood concentration at steady state

SECONDARY OUTCOMES:
AUC(0-τ)ss | Day 14 of each treatment period
  Area under the whole blood concentration curve during a dosage interval (τ=24 hours) at steady state
Cmax,ss | Day 14 of each treatment period
  Maximum whole blood concentration at steady state
Cmin,ss | Days 14 and 21 of each treatment period
  Minimum whole blood concentration at steady state
Cτ,ss | Days 14 and 21 of each treatment period
  Concentration at the end of the dosing interval at steady state
Cav | Days 14 and 21 of each treatment period
  Average concentration during a dosing interval: AUC(0-τ)/τ
Tmax,ss | Days 14 and 21 of each treatment period
  Time to reach maximum (peak) plasma concentration at steady state
AUC(0-τ)ss coefficient of variation | Days 14 and 21 of each treatment period
  Intra-patient pharmacokinetics variability evaluated by calculating AUC(0-τ)ss coefficient of variation
Cmax,ss coefficient of variation | Days 14 and 21 of each treatment period
  Intra-patient pharmacokinetics variability evaluated by calculating Cmax,ss coefficient of variation
% Fluctuation | Days 14 and 21 of each treatment period
  Degree of fluctuation of the analyte concentration levels over one dosing interval: 100*(Cmax,ss - Cmin,ss)/Cav.
%Swing | Days 14 and 21 of each treatment period
  Degree of change of the analyte concentration levels over one dosing interval: 100*(Cmax,ss - Cτ,ss)/Cτ,ss.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (13):
- France (7):
  - Sandoz Investigative Site, Grenoble
  - Sandoz Investigative Site, Limoges
  - Sandoz Investigative Site, Nantes
  - Sandoz Investigative Site, Strasbourg
  - Sandoz Investigative Site, Suresnes
  - Sandoz Investigative Site, Toulouse
  - Sandoz Investigative Site, Tours
- Germany (6):
  - Sandoz Investigative Site, Berlin
  - Sandoz Investigative Site, Bochum
  - Sandoz Investigative Site, Essen
  - Sandoz Investigative Site, Hanover
  - Sandoz Investigative Site, Kaiserslautern
  - Sandoz Investigative Site, Kiel

IPD SHARING:
Plan to Share IPD: No